CLINICAL TRIAL: NCT00558701
Title: Prospective, Randomized, Controlled Study of the Efficacy of a Silver-coated Nylon Dressing Plus Active or Sham Microcurrent for Healing Autogenous Skin Donor Sites
Brief Title: Microcurrent for Healing Autogenous Skin Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-07-003; I.2007.128 (Other: BAMC IRB)
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2015-08

CONDITIONS: Burns
Keywords: burns; donor site; healing; microcurrent
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microcurrent Stimulator + Silverlon (Active Comparator): Patients receiving active electrical stimulation (15-50 microamps) during treatment of skin donor sites with Silverlon wound contact dressing. Intervention is active electrical stimulation via microcurrent stimulator.
  Interventions: Device: Microcurrent stimulator; Device: Silverlon Wound Contact Dressing
- Silverlon alone (Sham Comparator): Patients receiving treatment of skin donor sites with Silverlon wound contact dressing alone (i.e., without active electrical stimulation)
  Interventions: Device: Silverlon Wound Contact Dressing

INTERVENTIONS:
Device: Microcurrent stimulator — Microcurrent stimulation from 15-50 microamps
  Arms: Microcurrent Stimulator + Silverlon
Device: Silverlon Wound Contact Dressing — Silver coated nylon dressing FDA approved for use on donor sites in burn patients

SUMMARY:
This single-center, prospective, randomized, and controlled study evaluated the efficacy of silver-coated dressing with active microcurrent in comparison to silver-coated dressing with sham microcurrent on wound-closure time for autogenous skin donor sites.

DETAILED DESCRIPTION:
The specific aims of the study are to evaluate the impact of active versus sham direct microcurrent application to silver nylon dressings in the treatment of donor sites for partial thickness thermal injuries. The primary endpoint is wound-closure time (re-epithelialization of 90% or more of wound surface). A secondary endpoint was infection. Exploratory assessments of clinical outcomes, including inflammation, and pain medication (type, dosage, route, timing) will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years of age
* burn less than 30% total body surface area
* burns not involving donor site area
* you need skin grafting to cover burns
* agree not to use other electronic devices that generate current during your study participation
* agree to come back for follow up visits at least every other day after discharge from hospital until donor site is healed

Exclusion Criteria:

* you have an illness that may affect how your wound heals such as diabetes, blood clotting disorder, cirrhosis, liver failure, peripheral vascular disease
* you are taking medications that could affect how your wound heals such as steroids, Plavix, Coumadin
* you have an infection of the skin or your bloodstream
* you are pregnant or nursing
* you are sensitive or allergic to silver or nylon
* your burn wounds are more than 30% of your total body surface area
* your site was previously harvested for grafting
* you have an implantable pacemaker device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo C Cancio, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- USAISR, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kauvar DS, Cancio LC, Wolf SE, Wade CE, Holcomb JB. Comparison of combat and non-combat burns from ongoing U.S. military operations. J Surg Res. 2006 May 15;132(2):195-200. doi: 10.1016/j.jss.2006.02.043. Epub 2006 Mar 31. PMID 16580688
- [Derived] Malin EW, Galin CM, Lairet KF, Huzar TF, Williams JF, Renz EM, Wolf SE, Cancio LC. Silver-coated nylon dressing plus active DC microcurrent for healing of autogenous skin donor sites. Ann Plast Surg. 2013 Nov;71(5):481-4. doi: 10.1097/SAP.0b013e31829d2311. PMID 23903090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microcurrent Stimulator + Silverlon | Silverlon Alone
Started | 15 | 15
Completed | 14 | 11
Not Completed | 1 | 4
Not completed — Protocol Deviations | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Microcurrent Stimulator + Silverlon: Patients receiving active electrical stimulation (15-50 microamps) during treatment of skin donor sites with Silverlon wound contact dressing.
  Intervention is active electrical stimulation via microcurrent stimulator.
  Microcurrent stimulator: Microcurrent stimulation from 15-50 microamps Silverlon Wound Contact Dressing: Silver coated nylon dressing FDA approved for use on donor sites in burn patients
- Total: Total of all reporting groups
Arm/Group | Microcurrent Stimulator + Silverlon | Silverlon Alone | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (9.5) | 33.8 (9.5) | 33.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Wound Healing
Description: Time to 90% confluent reepitheliazation of donor site, as indicator of wound healing
Time Frame: 20 days
Measure: Mean (Full Range); unit: days
Arm/Group | Microcurrent Stimulator + Silverlon | Silverlon Alone
Number analyzed (Participants) | 14 | 11
days | 10.8 [7 to 15] | 11.1 [8 to 14]

ADVERSE EVENTS:
Arm/Group | Microcurrent Stimulator + Silverlon | Silverlon Alone
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microcurrent Stimulator + Silverlon (N=14) | Silverlon Alone (N=11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — IRB found not to be attributable to study.
Deep Vein Thrombosis (DVT) (Vascular disorders) | 0 (0) | 1 (1) — Institutional Review Board (IRB) found not to be attributable to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes